CLINICAL TRIAL: NCT02120105
Title: Cystine Capacity Clinical Study (CysCap)
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 6402
Record Dates: First submitted 2013-06-04; First posted 2014-04-22 (Estimated); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Cystinuria
Keywords: Renal aminoaciduria; cystinuria; D-penicillamine; renal tubular transport; inborn errors; tiopronin; urolithiasis
MeSH Terms: conditions — Cystinuria; Renal Aminoacidurias; Urolithiasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cystinuria

SUMMARY:
The purpose of this study is to determine whether urinary cystine capacity, an assay used to measure the amount of cystine in the urine, can be used to predict stone recurrence in patients with cystinuria.

DETAILED DESCRIPTION:
Cystinuria is a rare genetic cause of kidney stones that leads to significant morbidity due to the recurrent nature of the disease. Despite recent advancements in knowledge about cystinuria, such as the discovery of the genetic defects that cause the disease, there have been very few studies of clinical determinants of recurrent stone formation. An optimal method of measuring cystine solubility in the urine has been lacking, and therefore response to pharmacologic and dietary therapy is often not known. Recently, a new assay to measure the amount of cystine in the urine was developed called Cystine Capacity, or CysCap. It is an assay that adds a pre-formed amount of cystine crystals to urine and measures the amount of cystine the urine can take up from the solid phase (in undersaturated urine) or gives up to solid phase (in supersaturated urine). This study seeks to examine how well this measure of urinary cystine predicts stone occurrence, with the ultimate goal of helping to guide therapy and preventing kidney stones in cystinurics.

This is an observational study over 3 years. Subjects who are enrolled in the study will perform semi-annual 24-hour urine collections. They will undergo imaging of the kidneys every 6 months to monitor kidney stone formation or growth, in order to correlate urinary parameters with clinical events. The study will examine how well the urinary cystine capacity predicts stone formation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed laboratory diagnosis of cystinuria will be included in this study. There will be no age barrier to inclusion, but included patients must be able to reliably collect urine for 24 hours. Men and women will be recruited equally and there are no restrictions for racial or ethnic origin in this study.
* Patient enrollment will require signing of an informed consent document approved by the Lenox Hill IRB.
* For children 8-18 years of age, signing an assent to participate will also be required.

Exclusion Criteria:

* Patients will be excluded if they cannot sign consent or assent.
* Furthermore if the patient cannot reliably collect urine for 24 hours or adhere to study follow up visit requirements.

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: For patients to be enrolled in this study they must have a diagnosis of cystinuria.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2017-02-24 (Actual); Study Completion 2017-02-24 (Actual)

PRIMARY OUTCOMES:
Cystine capacity will be correlated with recurrence or non-recurrence of stones | every 6 months over 3 years
  The primary end point will be cystine capacity in participants who do and do not have recurrence of stones seen on radiologic imaging in the ipsilateral kidney which was rendered stone-free prior to enrollment.
  Subjects who are enrolled in the study will perform semi-annual 24-hour urine collections for measurement of cystine capacity. They will undergo imaging of the kidneys every 6 months to monitor kidney stone formation or growth, in order to correlate urinary parameters with clinical events.

SECONDARY OUTCOMES:
24-hour urine cystine excretion | every 6 months over 3 years
  We will compare 24 hour urine cystine excretion in patients who remain stone free and those who experience stone recurrence.
episodes of renal colic and/or stone passage from a kidney that was previously stone-free | every 6 months over 3 years
  Assessed by renal imaging, either ultrasound or CT scan, every 6 months.
Evidence of new asymptomatic stones noted on the contralateral kidney | every 6 months over 3 year observational study
  Cystine capacity will be compared in participants with or without recurrence of stones in the contralateral kidney by renal ultrasound or CT scan

CONTACTS AND LOCATIONS:
Overall Officials: David S Goldfarb, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

REFERENCES:
- [Background] Goldfarb DS, Coe FL, Asplin JR. Urinary cystine excretion and capacity in patients with cystinuria. Kidney Int. 2006 Mar;69(6):1041-7. doi: 10.1038/sj.ki.5000104. PMID 16501494
- See also: Rare Kidney Stone Consortium — http://www.rarekidneystones.org/